CLINICAL TRIAL: NCT01485276
Title: Pilot Study of Bilateral Pedunculo-Pontine Nucleus (PPN) Deep Brain Stimulation for Patients With Parkinson Disease (PD) Who Have Persistent Gait Disturbance, Despite Bilateral Subthalamic Nucleus (STN) Deep Brain Stimulation
Brief Title: Combined Deep Brain Stimulation for Parkinson's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120012; 12-N-0012
Record Dates: First submitted 2011-12-02; First posted 2011-12-05 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2014-07-30

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation; Gait; Electrophysiology; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Procedure: DBS Surgery

SUMMARY:
Background:

- Deep brain stimulation (DBS) in the subthalamic nucleus (STN) is an approved treatment for Parkinson s disease. It stimulates a part of the brain that helps control symptoms like tremor, stiffness, and slow movements. However, many people continue to have unsteadiness and slowness while walking, trouble swallowing, and speech problems even with STN DBS. Another type of DBS focuses on a part of the brain called the pedunculopontine nucleus (PPN). PPN DBS has improved walking in some people with Parkinson's disease. Researchers want to see if combining the two types of DBS may help control symptoms better than STN DBS alone.

Objectives:

* To see if PPN DBS can help walking, balance, speaking, and swallowing in those who already have STN DBS.
* To study how the DBS combination affects brain function.

Eligibility:

- Individuals with Parkinson s disease who had STN DBS surgery at least 1 year ago, but still have difficulty walking, swallowing, and speaking.

Design:

* Participants will be screened with a physical exam and medical history. They will also have neurological tests and other tests to measure Parkinson s disease symptoms.
* This study requires eight visits over 1 year. One of the visits will be a 9- to 10-day admission to the NIH Clinical Center for DBS surgery.
* Participants will have PPN DBS surgery. The surgery will be done in two steps. In the first step, the leads will be placed in the brain. In the second step, 1 week later, the stimulator device will be placed in the chest or abdomen.
* One month after the surgery, participants will have a study visit to program the PPN DBS device to find settings that will improve walking and balance.
* Participants will have study visits 2, 3, 6, and 12 months after surgery. Each visit will be used to check the stimulators and make any adjustments needed to try to improve walking and balance or to lessen side effects. Participants will have tests of walking and balance, speech, and swallowing. Some tests will be done with different combinations of the stimulators on or off to see the effects of each set of stimulators.

DETAILED DESCRIPTION:
OBJECTIVE:

1. Determine if bilateral Pedunculo-Pontine Nucleus (PPN) Deep Brain Stimulation (DBS) will improve gait and balance problems in Parkinson Disease (PD) patients whose other disease features have responded to bilateral subthalamic nucleus (STN) DBS and medications
2. Determine if bilateral PPN DBS will improve swallowing function in Parkinson Disease patients treated with bilateral STN DBS and medication
3. Obtain electrophysiological data related to PPN
4. Obtain data related to the physiological relationship of the STN and PPN

STUDY POPULATION:

Three (3) subjects with clinically diagnosed PD who have undergone bilateral STN DBS at least one year prior to enrollment, who continue to have gait and balance disturbance.

DESIGN:

Pilot study of 3 patients with clinically diagnosed PD who have undergone bilateral STN DBS at least one year prior to enrollment. Baseline evaluation will include neurologic clinical evaluation, postural and gait physiologic and clinical assessment, brain imaging, and video swallow evaluation. The patients will undergo the surgical procedure (bilateral PPN DBS implant) in the Clinical Center (CC). Electrode recordings will be obtained from the implant site within the first week post-operatively from an externalized lead, then the second surgical stage (pulse generator implant) will take place, also in the Clinical Center. The patients will undergo programming to optimal parameters and appropriate follow-up, and the outcome measures will be assessed at 1 week and 1, 3, 6 and 12 months post-surgery. Recruitment will be staggered and at least 4 weeks will be required between different patients beginning the study. Recruitment will be halted if major unexpected side-effects occur causing concern about the welfare of patients.

This study is to serve as the basis for an extended, larger study, which would be properly powered to answer the clinical research questions. The efficacy criterion for translation into a larger study will be 30% improvement in the primary outcome in 2 out of the 3 patients. In addition, we will obtain valuable and for the most part novel data regarding the electrophysiologic properties of the PPN and the complex interactions between basal ganglia (BG) components in the parkinsonian state and the response to DBS. The data obtained in this study will inform the design, selection and treatment paradigms in future larger studies.

OUTCOME MEASURES:

Primary:

* Change in the amount of time needed to complete a standardized timed up and go (TUG) study at 6 months post-surgery on stimulation
* Change in the amount of time needed to complete a standardized timed up and go (TUG) study at 6 months post-surgery on stimulation, compared to off stimulation.

Secondary:

* Change in time needed to complete the TUG study at 1, 3 and 12 months post-surgery on stimulation
* UPDRS part III score and UPDRS part III points 27-30 at 1, 3, 6 and 12 months on stimulation
* Parkinson's Disease Questionnaire (PDQ 31) quality of life questionnaire at 6 months
* Change in static and dynamic posturography outcome parameters at 1, 3, 6 and 12 months on stimulation
* Number of adverse events during the follow-up period
* Change in timed and non-timed variables of swallowing function at 6 months
* Recorded physiologic function of PPN with STN stimulator off and on at rest and during gait
* Changes in the patient global impression of change at 1, 3, 6, and 12 months. All the outcome measures are assessed on best medical therapy..

ELIGIBILITY:
-INCLUSION CRITERIA:

i. Greater than 22 years of age

ii. Successful bilateral STN DBS implants for at least 1 year

iii. At least 30% improvement in the motor UPDRS following STN therapy, by history and record review

iv. Improved UPDRS and self assessment questionnaire following STN DBS by at least 20%, by history and record review.

v. Good STN DBS placement assessed with imaging (CT scan, MRI or fused CT-MRI imaging)

vii. Persistent gait disturbance as ascertained by abnormal performance on the time-up-and-go test compared to age-matched controls as well as preoperative evaluation with posturography and quantitative gait assessment (values compared to normal age-matched controls) at least 30% difference from age-matched controls on either measure.

vii. Persistent speech and swallowing problems as measured by a minimum score of I in items 5 and 7 of the UPDRS

viii. Evaluation by an independent movement disorders specialist who will confirm gait disturbance in the presence of STN stimulation.

EXCLUSION CRITERIA:

i. Pregnant or nursing women

ii. Cognitively impaired subjects as determined by pre-operative neuropsychology evaluation, including Mattis Dementia Rating Scale (DRS). Patients scoring below 70 on the Mattis DRS will be excluded.

iii. Depressed subjects as determined by the neuropsychology screen, including Beck Depression Inventory. Patients scoring above 20 on the Beck inventory will be excluded.

iv. Patients with uncontrolled co-existing medical conditions: uncontrolled systemic hypertension with values above 170/100; heart disease needing intervention; respiratory disease needing intervention; uncorrected coagulation abnormalities or need for therapeutic anticoagulation which cannot be interrupted; any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.

v. Patients with metal objects in their body that are not MRI compatible, excluding the previous STN DBS hardware

vi. Patients who have a history of seizures, require repeated magnetic resonance imaging (MRI) scans or have had a cranial neurosurgical procedure since receiving an STN implant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11-08; Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
Change in the amount of time needed to complete a standardized timed up and go (TUG) study at 6 months post-surgery on stimulation

SECONDARY OUTCOMES:
TUG study at 1, 3 and 12 months post-surgery.
UPDRS III score and UPDRS III points 27-30 at 1, 3, 6 and 12 months
PDQ 31 questionnaire at 6 months
Swallowing function at 6 moths
Static and dynamic posturography parameters at 1, 3, 6 and 12 months on stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Rodriguez-Oroz MC, Obeso JA, Lang AE, Houeto JL, Pollak P, Rehncrona S, Kulisevsky J, Albanese A, Volkmann J, Hariz MI, Quinn NP, Speelman JD, Guridi J, Zamarbide I, Gironell A, Molet J, Pascual-Sedano B, Pidoux B, Bonnet AM, Agid Y, Xie J, Benabid AL, Lozano AM, Saint-Cyr J, Romito L, Contarino MF, Scerrati M, Fraix V, Van Blercom N. Bilateral deep brain stimulation in Parkinson's disease: a multicentre study with 4 years follow-up. Brain. 2005 Oct;128(Pt 10):2240-9. doi: 10.1093/brain/awh571. Epub 2005 Jun 23. PMID 15975946
- [Background] Benabid AL, Pollak P, Gross C, Hoffmann D, Benazzouz A, Gao DM, Laurent A, Gentil M, Perret J. Acute and long-term effects of subthalamic nucleus stimulation in Parkinson's disease. Stereotact Funct Neurosurg. 1994;62(1-4):76-84. doi: 10.1159/000098600. PMID 7631092
- [Background] Kleiner-Fisman G, Fisman DN, Sime E, Saint-Cyr JA, Lozano AM, Lang AE. Long-term follow up of bilateral deep brain stimulation of the subthalamic nucleus in patients with advanced Parkinson disease. J Neurosurg. 2003 Sep;99(3):489-95. doi: 10.3171/jns.2003.99.3.0489. PMID 12959435